CLINICAL TRIAL: NCT00773851
Title: Mesh Shrinkage Following Transfacial Suturing Versus Stapler for Mesh Fixation in Laparoscopic Ventral Hernia Repair: a Prospective, Randomised Blinded Study
Brief Title: Transfacial Sutures Versus Stapler for Mesh Fixation in Laparoscopic Ventral Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Collaborators: Sofradim Production (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KEK_11/05
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Ventral Hernia; Pain
Keywords: ventral hernia; laparoscopy; mesh; recurrence
MeSH Terms: conditions — Hernia, Ventral; Pain; Recurrence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other): transfacial sutures
  Interventions: Procedure: mesh fixation by transfacial sutures
- B (Other): staples
  Interventions: Procedure: mesh fixation by staples

INTERVENTIONS:
Procedure: mesh fixation by transfacial sutures — mesh fixation by transfacial sutures
  Arms: A
Procedure: mesh fixation by staples — mesh fixation by staples
  Arms: B

SUMMARY:
Hernia of the abdominal wall occur frequently after various surgical procedures of the abdomen and are increasingly performed by laparoscopic means. Different mesh fixation techniques are applied, but the influence of mesh fixation on shrinkage is not known in human patients. Therefore, mesh shrinkage was assessed using two different techniques for fixation.

DETAILED DESCRIPTION:
Ventral hernia repair is increasingly performed by laparoscopic means. While mesh ingrowth and shrink-age has been analysed in the experimental setting, there is scarce data available in humans. In addition, different mesh fixation techniques are applied, but the influence of mesh fixation on shrinkage is not known in human patients.

Mesh shrinkage is assessed using two different techniques for fixation.

Blinded randomized trial using a Parietene composite mesh for laparoscopic ventral hernia repair. Patients with ventral hernias of no larger than 8 cm were assigned to either mesh fixation using transfacial nonabsorbable sutures or titan tacks. Primary endpoint was mesh migration, secondary endpoints were mesh shrinkage, surgical morbidity and pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with incisional hernia smaller than 8cm in diameter
* obtained informed consent

Exclusion Criteria:

* Pregnancy
* Residual intraperitoneal mesh
* contaminated abdominal cavity
* longterm use of corticosteroids and other immunosuppressive agents
* bodymass index > 45
* general contradictions for laparoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-04; Primary Completion 2008-02 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
mesh shrinkage | perioperative, 6 weeks, 6 months postoperative

SECONDARY OUTCOMES:
mesh dislocation | perioperative, 6 weeks postoperative,6 months postoperative
pain | perioperative, 6 weeks postoperative,6 months, 12 moths postoperative
recurrence | perioperative, 6 weeks postoperative,6 months, 12 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Guido1 Beldi, MD, Principal Investigator — Bern University Hospital
Locations (1):
- Dep. of Visceral and Transplantsurgery, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Heniford BT, Park A, Ramshaw BJ, Voeller G. Laparoscopic repair of ventral hernias: nine years' experience with 850 consecutive hernias. Ann Surg. 2003 Sep;238(3):391-9; discussion 399-400. doi: 10.1097/01.sla.0000086662.49499.ab. PMID 14501505
- [Background] Borrazzo EC, Belmont MF, Boffa D, Fowler DL. Effect of prosthetic material on adhesion formation after laparoscopic ventral hernia repair in a porcine model. Hernia. 2004 May;8(2):108-12. doi: 10.1007/s10029-003-0181-6. Epub 2003 Nov 21. PMID 14634842
- [Background] van't Riet M, de Vos van Steenwijk PJ, Kleinrensink GJ, Steyerberg EW, Bonjer HJ. Tensile strength of mesh fixation methods in laparoscopic incisional hernia repair. Surg Endosc. 2002 Dec;16(12):1713-6. doi: 10.1007/s00464-001-9202-7. Epub 2002 Jul 8. PMID 12098028
- [Background] Winslow ER, Diaz S, Desai K, Meininger T, Soper NJ, Klingensmith ME. Laparoscopic incisional hernia repair in a porcine model: what do transfixion sutures add? Surg Endosc. 2004 Mar;18(3):529-35. doi: 10.1007/s00464-003-8519-9. Epub 2004 Feb 2. PMID 14752650
- [Background] LeBlanc KA. The critical technical aspects of laparoscopic repair of ventral and incisional hernias. Am Surg. 2001 Aug;67(8):809-12. PMID 11510590
- [Background] Carbajo MA, Martp del Olmo JC, Blanco JI, Toledano M, de la Cuesta C, Ferreras C, Vaquero C. Laparoscopic approach to incisional hernia. Surg Endosc. 2003 Jan;17(1):118-22. doi: 10.1007/s00464-002-9079-0. Epub 2002 Oct 29. PMID 12399849
- [Background] Chelala E, Gaede F, Douillez V, Dessily M, Alle JL. The suturing concept for laparoscopic mesh fixation in ventral and incisional hernias: preliminary results. Hernia. 2003 Dec;7(4):191-6. doi: 10.1007/s10029-003-0143-z. Epub 2003 Jun 13. PMID 12811619
- [Background] LeBlanc KA. Tack hernia: a new entity. JSLS. 2003 Oct-Dec;7(4):383-7. PMID 14626408
- [Background] Leber GE, Garb JL, Alexander AI, Reed WP. Long-term complications associated with prosthetic repair of incisional hernias. Arch Surg. 1998 Apr;133(4):378-82. doi: 10.1001/archsurg.133.4.378. PMID 9565117
- [Background] Schumpelick V, Klinge U. Prosthetic implants for hernia repair. Br J Surg. 2003 Dec;90(12):1457-8. doi: 10.1002/bjs.4385. No abstract available. PMID 14648721